CLINICAL TRIAL: NCT00805935
Title: A Multi-Center, Randomized, Open-Label Evaluation of MENOPUR® Versus FOLLISTIM® in Polycystic Ovarian Syndrome (PCOS) Patients
Brief Title: Menopur® Versus Follistim® in Polycystic Ovarian Syndrome (PCOS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-05
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Results first posted 2012-01-25 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2012-01

CONDITIONS: Polycystic Ovarian Syndrome; Infertility
Keywords: pre-menopausal women; PCOS; polycystic ovarian syndrome; infertility; IVF; in vitro fertilization
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Menotropins; Progesterone; follitropin beta; Oils; Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Menotropin/Progesterone vaginal insert (Experimental): Highly purified menotropin (Menopur®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone vaginal insert (Endometrin®) 100 mg starts on the day following oocyte retrieval and continues for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Menotropin; Drug: Progesterone vaginal insert; Drug: leuprolide acetate
- Menotropin/Progesterone in oil (Experimental): Menotropin (Menopur®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in oil 50 mg injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Menotropin; Drug: Progesterone in oil; Drug: leuprolide acetate
- Follitropin beta/Progesterone vaginal insert (Active Comparator): Follitropin beta (Follistim Pen®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone vaginal insert (Endometrin®) 50 mg injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Progesterone vaginal insert; Drug: Follitropin beta; Drug: leuprolide acetate
- Follitropin beta/Progesterone in oil (Active Comparator): Follitropin beta (Follistim Pen®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in oil 50 mg injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
  Interventions: Drug: Follitropin beta; Drug: Progesterone in oil; Drug: leuprolide acetate

INTERVENTIONS:
Drug: Menotropin — 225 IU (up to 450 IU) by subcutaneous injection once per day for up to about 15 days.
  Other Names: Menopur®
  Arms: Menotropin/Progesterone in oil; Menotropin/Progesterone vaginal insert
Drug: Progesterone vaginal insert — 100 mg inserted vaginally 2 or 3 times daily (BID or TID) (start on the day after oocyte retrieval) until 10 weeks gestation or confirmation of negative pregnancy test.
  Other Names: Endometrin®
  Arms: Follitropin beta/Progesterone vaginal insert; Menotropin/Progesterone vaginal insert
Drug: Follitropin beta — 225 IU (up to 450 IU) by subcutaneous injection once per day for up to about 15 days.
  Other Names: Follistim Pen®
  Arms: Follitropin beta/Progesterone in oil; Follitropin beta/Progesterone vaginal insert
Drug: Progesterone in oil — 50 mg by intramuscular injection once per day, starting on the day after oocyte retrieval until 10 weeks gestation or confirmation of negative pregnancy test.
  Arms: Follitropin beta/Progesterone in oil; Menotropin/Progesterone in oil
Drug: leuprolide acetate — Daily administration of 0.5mg of leuprolide acetate (depot formulations were not permitted) began on Day 21 following onset of menses, and then decreased to 0.25 mg when gonadotropin therapy was initiated.
  Other Names: Lupron

SUMMARY:
This multicenter, randomized, open-label exploratory study will be performed in approximately 200 polycystic ovary syndrome (PCOS) but otherwise healthy females undergoing in vitro fertilization (IVF). Each study center will follow its standard practice for in vitro fertilization (IVF) within the study parameters as noted in this protocol. The study centers will use marketed products purchased from Schraft's Pharmacy for all phases of the study (down-regulation, stimulation, ovulation induction, and luteal support). Subjects will be randomly assigned to highly purified menotropin (Menopur®) or follitropin beta (Follistim Pen®) for stimulation and progesterone vaginal insert (Endometrin®) or progesterone in oil for luteal support. Subjects will return to the study center for regular scheduled clinic visits as required per in vitro fertilization (IVF) protocol at the site and at specified times during the cycle (Stimulation Day 6, Day of human chorionic gonadotropin (hCG), and first serum pregnancy test) for estradiol (E2), progesterone (P4) and human chorionic gonadotropin (hCG) labs. All subjects will be required to complete a final study visit at completion of luteal support or negative serum pregnancy test following embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal females between the ages of 18 and 42 years
2. Diagnosed with polycystic ovary syndrome (PCOS), using criteria adopted as the 2003 Rotterdam PCOS Consensus (2 out of 3, excluding other etiologies [congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome])

   * Oligo- or anovulation
   * Clinical and/or biochemical signs of hyperandrogenism
   * Polycystic ovaries
3. Body mass index (BMI) of 18-39
4. Early follicular phase (Day 3) follicle stimulating hormone (FSH) < 15 IU/L and estradiol (E2) within normal limits
5. Documented history of infertility (e.g., unable to conceive for at least one year, or for 6 months for women > 38 years of age, or bilateral tubal occlusion or absence, or male factor but excluding severe male factor requiring invasive or surgical sperm retrieval. Donor sperm may be used.)
6. Transvaginal ultrasound at screening consistent with findings adequate for assisted reproductive technology (ART) with respect to uterus and adnexa
7. Signed informed consent

Exclusion Criteria:

1. Gestational or surrogate carrier, donor oocyte
2. Presence of any clinically relevant systemic disease (e.g., uncontrolled thyroid or adrenal dysfunction, an organic intracranial lesion such as a pituitary tumor, insulin-dependent diabetes mellitus, uterine cancer)
3. Surgical or medical condition which, in the judgment of the Investigator or Sponsor, may interfere with absorption, distribution, metabolism, or excretion of the drugs to be used
4. Two or more previous failed in vitro fertilization (IVF) cycles or in vitro fertilization (IVF)/assisted reproductive technology (ART) failure due to a poor response to gonadotropins, defined as development of 2 mature follicles
5. History of recurrent pregnancy loss, defined as more than two clinical losses
6. Presence of abnormal uterine bleeding of undetermined origin
7. Current or recent substance abuse, including alcohol or smoking > 10 cigarettes per day
8. Refusal or inability to comply with the requirements of the Protocol for any reason, including scheduled clinic visits and laboratory tests
9. Participation in any experimental drug study within 30 days prior to Screening
10. Severe male factor requiring invasive or surgical sperm retrieval (e.g., microsurgical epididymal sperm aspiration [MESA], testicular sperm extraction [TESE])
11. Prior hypersensitivity to any of the protocol drugs

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (6):
- United States (6):
  - Conceptions Reproductive Associates of Colorado, Littleton, Colorado
  - Women's Medical Research Group LLC, Florida, Clearwater, Florida
  - Fertility Center of Illinois, Chicago, Illinois
  - Weill Cornell Medical College, New York, New York
  - Women & Infants' Hospital of RI, Providence, Rhode Island
  - Center for Assisted Reproduction, Bedford, Texas

REFERENCES:
- [Derived] Beltsos AN, Sanchez MD, Doody KJ, Bush MR, Domar AD, Collins MG. Patients' administration preferences: progesterone vaginal insert (Endometrin(R)) compared to intramuscular progesterone for Luteal phase support. Reprod Health. 2014 Nov 11;11:78. doi: 10.1186/1742-4755-11-78. PMID 25385669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The original plan was for 200 participants to be enrolled across six (6) women's reproductive study centers across the US.
Pre-assignment Details: 127 patients were screened. 120 patients were randomized. Of the randomized patients, 10 did not receive treatment. 110 randomized participants started the study on treatment.
Groups:
- Menotropin/Progesterone in Oil: Highly purified menotropin (Menopur®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in oil 50 mg injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
- Follitropin Beta/Progesterone Vaginal Insert: Follitropin beta (Follistim®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone vaginal insert (Endometrin®) 50 mg injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
- Follitropin Beta/Progesterone in Oil: Follitropin beta (Follistim®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  Progesterone in oil 50 mg injections start on the day following oocyte retrieval and continue for a total duration of 10 weeks or until a negative pregnancy test is obtained.
Period: Overall Study
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Started | 25 | 27 | 28 | 30
Completed | 12 | 8 | 13 | 19
Not Completed | 13 | 19 | 15 | 11
Not completed — Stimulation Failure | 1 | 5 | 2 | 2
Not completed — Cycle cancelled | 0 | 0 | 2 | 0
Not completed — Cycle cancellation for risk of OHSS | 1 | 0 | 1 | 0
Not completed — Ovarian hyperstimulation syndrome(OHSS) | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — No positive serum pregnancy | 8 | 7 | 6 | 5
Not completed — Pregnancy not confirmed by ultrasound | 0 | 0 | 0 | 1
Not completed — Pregnancy loss/miscarriage | 2 | 0 | 0 | 0
Not completed — Biochemical pregnancy | 0 | 1 | 0 | 0
Not completed — Chemical pregnancy | 0 | 5 | 3 | 2
Not completed — Ectopic pregnancy | 0 | 0 | 1 | 0
Not completed — Serious Adverse Event-congenital anomaly | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil | Total
Number analyzed (Participants) | 25 | 27 | 28 | 30 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 27 | 28 | 30 | 110
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 28 | 30 | 110
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 18 | 18 | 20 | 25 | 81
  African American | 0 | 1 | 0 | 0 | 1
  Asian | 5 | 1 | 4 | 1 | 11
  Hispanic | 2 | 7 | 4 | 3 | 16
  Other | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With Cycle Cancellation Due to Risk of Ovarian Hyperstimulation Syndrome (OHSS) Between Weeks 1 - 3
Description: A count of participants whose discontinuation was clearly documented on the study completion/termination form as cycle cancellation for risk of ovarian hyperstimulation syndrome (OHSS).
Time Frame: weeks 1-3
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
Participants
  Yes | 1 | 0 | 1 | 0
  No | 24 | 27 | 27 | 30
Statistical Analysis 1: Comparison: Menotropin/Progesterone Vaginal Insert vs Follitropin Beta/Progesterone Vaginal Insert; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: Menotropin/Progesterone in Oil vs Follitropin Beta/Progesterone in Oil; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Menotropin/Progesterone Vaginal Insert vs Menotropin/Progesterone in Oil; Comparing Progesterone vaginal insert to Progesterone in oil within the menotropin treatments arms; Test type: Superiority or Other; p = 0.481, Fisher Exact
Statistical Analysis 4: Comparison: Follitropin Beta/Progesterone Vaginal Insert vs Follitropin Beta/Progesterone in Oil; Comparing Progesterone vaginal insert to Progesterone in oil within the follitropin beta treatment group; Test type: Superiority or Other; p = 0.483, Fisher Exact

2. Secondary Outcome: Number of Follicles Observed at Day 15
Description: The mean number of follicles observed in both ovaries at the last transvaginal ultrasound in the stimulation phase.
Time Frame: approximately day 15
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Follicles
Groups:
- Menotropin: Highly purified menotropin (Menopur®) 225 IU by subcutaneous injection once per day from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  This group combines the two treatment arms that use Highly purified menotropin (Menopur®) for ovarian stimulation. This treatment is followed by luteal support using either Progesterone vaginal insert (Endometrin®) or progesterone in oil.
- Follitropin Beta: Follitropin beta (Follistim®) 225 IU from day 1-6 of menstrual cycle. May be adjusted up to 450 IU daily for more days until human chorionic gonadotropin (hCG) criteria are met.
  This group combines the two treatment arms that use Follitropin beta (Follistim®) for ovarian stimulation. This treatment is followed by luteal support using either Progesterone vaginal insert (Endometrin®) or progesterone in oil.
Arm/Group | Menotropin | Follitropin Beta
Number analyzed (Participants) | 52 | 58
Follicles | 27.7 (12.8) | 30.5 (16.1)

3. Secondary Outcome: Number of Oocytes Retrieved at Day 18
Description: The mean number of oocytes retrieved approximately 36 hours after hCG (Novarel®) administration and fertilized (by insemination or intra cytoplasmic sperm injection (ICSI)) according to site-specific procedures.
Time Frame: approximately day 18
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Oocytes
Arm/Group | Menotropin | Follitropin Beta
Number analyzed (Participants) | 52 | 58
Oocytes | 13.0 (7.7) | 15.6 (8.6)

4. Secondary Outcome: Percentage of Oocytes Fertilized of the Total Number of Oocytes Retrieved
Description: The fertilization rate for each participant was the percentage of the number of oocytes inseminated of the total number of oocytes retrieved.
Time Frame: approximately day 19
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of oocytes retrieved
Arm/Group | Menotropin | Follitropin Beta
Number analyzed (Participants) | 52 | 58
Percentage of oocytes retrieved | 17.1 | 24.8

5. Secondary Outcome: Number of Embryos Transferred at Three Stages of Development Before Implantation
Description: The number of embryos, morulas and blastocysts transferred to the study participant on either day 3 or day 5 following fertilization. Embryos represent the earliest development stage and contain 2-8 cells.
  Morulas, the next stage, continued cellular cleavage results in a 16-30 cell solid sphere. Morula further develop into blastocyst, which contains 70-100 cells in a hollow spherical shape.
Time Frame: approximately day 24
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Embryos
Arm/Group | Menotropin | Follitropin Beta
Number analyzed (Participants) | 52 | 58
Embryos
  Number of embryos transferred | 2.0 (0.7) | 2.0 (0.5)
  Number of morula transferred | 0.0 (0.1) | 0.1 (0.4)
  Number of blastocyst transferred | 0.8 (0.9) | 1.1 (0.9)

6. Secondary Outcome: Number of Embryos Frozen
Description: The number of embryos that were not transferred but instead were frozen for future use.
Time Frame: approximately day 24
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Embryos
Arm/Group | Menotropin | Follitropin Beta
Number analyzed (Participants) | 52 | 58
Embryos | 1.9 (2.3) | 1.9 (2.6)

7. Secondary Outcome: Percentage of Participants With Biochemical Pregnancy at Approximately Day 38
Description: Biochemical pregnancy is a positive β-hCG pregnancy test 12-14 days post embryo transfer.
Time Frame: approximately day 38 (Day 14 post embryo transfer)
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
Percentage of participants | 60.0 | 55.6 | 60.7 | 73.3

8. Secondary Outcome: Percentage of Participants With Clinical Pregnancy at Week 7
Description: Clinical pregnancy is the confirmation of the presence of intrauterine gestational sacs on pregnancy ultrasound examination.
Time Frame: approximately Day 52
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
Percentage of participants | 56.0 | 33.3 | 46.4 | 66.7

9. Secondary Outcome: Percentage of Participants With Ongoing Pregnancy at Week 9
Description: as for outcome 8
Time Frame: approximately Day 65
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
Percentage of participants | 48.0 | 33.3 | 46.4 | 63.3

10. Secondary Outcome: Estradiol Levels at Day 6
Description: Estradiol monitoring during fertility therapy assesses follicular growth and is useful in monitoring the treatment. Blood tests sent to a central laboratory to obtain estradiol levels.
Time Frame: Day 6
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
pg/mL | 354.6 (331.3) | 268.2 (260.7) | 617.5 (409.6) | 550.5 (486.9)

11. Secondary Outcome: Human Chorionic Gonadotropin (hCG) Levels at Day 6
Description: Blood tests were sent to a central laboratory to obtain hCG levels.
Time Frame: Day 6
Population: Intend-to-treat (ITT) population -- all randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: mIU/ml
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
mIU/ml | 1.0 (0.2) | 1.0 (0.0) | 1.0 (0.0) | 1.0 (0.0)

12. Secondary Outcome: Progesterone Levels at Human Chorionic Gonadotropin (hCG) Administration
Description: Blood tests were sent to a central laboratory to obtain progesterone levels.
Time Frame: approximately day 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 23 | 21 | 23 | 28
ng/mL | 1.3 (0.7) | 1.1 (0.4) | 1.7 (0.9) | 1.3 (0.6)

13. Secondary Outcome: Number of Live Births Resulting From the In Vitro Fertilization Process
Description: Number of live births resulting from the IVF process
Time Frame: Approximately 10 months
Population: Database was locked prior to most participants giving birth.
Measure: Number; unit: Live births
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Participants With Treatment Emergent Adverse Events
Description: Number of participants with adverse events (AEs) that started after first treatment. Severity used a three point scale:
  mild=awareness of signs/symptoms, but no disruption of usual activity moderate=event sufficient to affect usual activity (disturbing) severe=event causes inability to work or perform usual activities (unacceptable) Relatedness to study treatment used a four point scale: unrelated, unlikely, possible, probable.
  Seriousness refers to death, hospitalization, a life-threatening experience, persistent or significant disability/incapacity, or congenital anomaly.
Time Frame: Week 1 to week12
Population: Safety population all randomized and treated participants. The safety population is identical intent-to- treat (ITT) population in this study
Measure: Number; unit: Participants
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Number analyzed (Participants) | 25 | 27 | 28 | 30
Participants
  With at least one adverse event | 9 | 12 | 15 | 14
  With at least one mild or moderate adverse event | 9 | 11 | 15 | 14
  With at least one severe adverse event | 0 | 2 | 1 | 0
  With at least one serious adverse event | 0 | 1 | 0 | 0
  With at least one unrelated or unlikely AE | 8 | 11 | 12 | 13
  With at least one possibly or probably related AE | 3 | 7 | 8 | 6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from Day 1 to Week 12.
Description: Multiple events in the same system organ class for a subject are only counted once for that system organ class.
Arm/Group | Menotropin/Progesterone Vaginal Insert | Menotropin/Progesterone in Oil | Follitropin Beta/Progesterone Vaginal Insert | Follitropin Beta/Progesterone in Oil
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/27 | 0/28 | 0/30
Other Adverse Events (participants affected / at risk) | 9/25 | 11/27 | 15/28 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menotropin/Progesterone Vaginal Insert (N=25) | Menotropin/Progesterone in Oil (N=27) | Follitropin Beta/Progesterone Vaginal Insert (N=28) | Follitropin Beta/Progesterone in Oil (N=30)
Conjoined Twins (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menotropin/Progesterone Vaginal Insert (N=25) | Menotropin/Progesterone in Oil (N=27) | Follitropin Beta/Progesterone Vaginal Insert (N=28) | Follitropin Beta/Progesterone in Oil (N=30)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 3
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Injection site anaesthesia (General disorders) | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 1
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 | 3 | 3 | 3
Procedural pain (Injury, poisoning and procedural complications) | 4 | 5 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 2
Antepartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian hyperstimulation (Reproductive system and breast disorders) | 2 | 2 | 2 | 2
Pelvic Discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine Spasm (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hot flush (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.